CLINICAL TRIAL: NCT06812026
Title: Comparison of the Effects of Melatonin and Lymphatic Drainage Massage on Pain, Edema, and Mouth Opening Following Impacted Third Molar Extraction
Brief Title: Effects of Melatonin and Massage After Third Molar Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: E.173684
Record Dates: First submitted 2025-01-27; First posted 2025-02-06 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Melatonin
Keywords: edema; tooth removal; melatonin
MeSH Terms: conditions — Edema | interventions — Massage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- control: during the postoperative period receive any lymphatic drainage massage and melatonin
  Interventions: Other: no melatonin and massage
- study melatonin: during the postoperative period receive only melatonin pills
  Interventions: Dietary Supplement: receive melatonin
- study lymphatic drainage massage: during the postoperative period receive only lymphatic drainage massage
  Interventions: Other: receiving lymphatic drainage

INTERVENTIONS:
Other: no melatonin and massage — receiving no melatonin and massage
  Groups: control
Dietary Supplement: receive melatonin — receiving only melatıonin pills
  Groups: study melatonin
Other: receiving lymphatic drainage — receiving lymphatic drainage massage
  Groups: study lymphatic drainage massage

SUMMARY:
Lymphatic drainage massage is an important practice, especially for reducing edema. It is a very gentle, monotonous, slow, rhythmic massage applied to the skin surface. It accelerates the flow of lymph fluid and provides comfort by minimizing swelling. Lymphatic drainage massage, which is frequently used after impacted third molar surgery, helps reduce edema and increases patient comfort during the postoperative period.

Melatonin, a hormone produced by the pineal gland, is a neurochemical substance that works in harmony with the body's natural rhythm. In addition to the brain, it is found in the retina, bone marrow, intestines, skin, and various blood cells. Conditions such as insomnia or jet lag may benefit from melatonin supplements. Besides contributing to sleep quality, melatonin may also assist in regulating the immune system, body temperature, blood pressure, and cortisol hormone levels.

DETAILED DESCRIPTION:
Another important function of melatonin is that it is a very powerful free radical scavenger. Melatonin can neutralize both reactive oxygen species and reactive nitrogen species. It is also known to capture highly toxic hydroxyl radicals, peroxynitrite anions, and peroxyl radicals. In some cases, melatonin inhibits nitric oxide synthase, a prooxidant enzyme. Additionally, it stimulates the mRNA levels of superoxide dismutase enzyme and is known to activate glutathione peroxidase, glutathione reductase, and glucose-6-phosphate dehydrogenase. After reacting with the hydroxyl free radical (OH•), melatonin transforms into an indolyl cation radical, which is noted to capture the superoxide radical (O2 · -) in the environment and exhibit antioxidant activity. Due to this powerful antioxidant property, its effects on pain and edema have been investigated in some studies. In these studies, pre-op/post-op melatonin application has been shown to reduce postoperative pain and accelerate sensory healing due to melatonin's antioxidant effects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients need for removal surgery of impacted third molars.
2. Patients without systemic diseases.

Exclusion Criteria:

1. Presence of systemic diseases affecting general health.
2. Presence of a malignant disease in the head and neck region.
3. Patients with any bleeding disorders.
4. Patients with cardiovascular diseases or those undergoing anticoagulant or antiplatelet therapy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: who need impacted tooth removal surgery in the rutine clinic patients
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-10 (Estimated)

PRIMARY OUTCOMES:
melatonin effect on edema: Postoperative edema will be measured preoperatively and on the 3rd and 7th days. Distances between the gonion-lateral canthus and tragus-labial commissure will be measured and recorded with a thread. | postoperative 7 days
  during the post operative periods patients receive melatonin pill until 7 days

SECONDARY OUTCOMES:
Lymphatic drainage massage effect on edema: Postoperative edema will be measured preoperatively and on the 3rd and 7th days. Distances between the gonion-lateral canthus and tragus-labial commissure will be measured and recorded with a thread. | postoperative 7 days
  during the post operative periods patients receive lymphatic drainage massage until 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf Universty, Istanbul, Fatih, Turkey (Türkiye)